CLINICAL TRIAL: NCT00940888
Title: SJ4 Post Approval Study
Brief Title: SJ4 Post Approval Study in Implantable Cardioverter-Defibrillator and Cardiac Resynchronization Therapy Defibrillator Patients
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: 60020938
Record Dates: First submitted 2009-07-14; First posted 2009-07-16 (Estimated); Results first posted 2017-08-14 (Actual); Last update posted 2019-02-04 (Actual); Status verified 2019-01

CONDITIONS: Tachyarrhythmias; Sudden Cardiac Death; Heart Failure
Keywords: ICD; CRTD; Heart Failure; DF4
MeSH Terms: conditions — Tachycardia; Death, Sudden, Cardiac; Heart Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- No treatment: ICD/CRTD-indicated
  Interventions: Device: SJ4 connector and RV high voltage SJ4 lead

INTERVENTIONS:
Device: SJ4 connector and RV high voltage SJ4 lead — Standard of care implantation of SJ4 device system

SUMMARY:
The purpose of this study is to characterize the chronic performance of the St. Jude Medical SJ4 connector and RV high voltage SJ4 leads.

ELIGIBILITY:
Inclusion Criteria:

* Have an approved indication per ACC/AHA/HRS guidelines for implantation of heart failure or life-threatening ventricular tachyarrhythmias and will be implanted with a St. Jude Medical SJ4 system.
* Have the ability to provide informed consent for study participating and be willing and able to comply with the prescribed follow-up test and schedule of evaluations.

Exclusion Criteria:

* Be currently participating in a clinical investigation that includes an active treatment arm.
* Have a life expectancy of less than 6 months due to any condition.
* Be less than 18 years of age.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ICD and CRTD indicated patients
Sampling Method: Non-Probability Sample
Enrollment: 1701 (Actual)
Dates: Start 2009-06; Primary Completion 2015-09 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Wilkoff, MD, Principal Investigator — The Clevleland Clinic Foundation
Locations (1):
- The Cleveland Clinic Foundation, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- SJ4 System Implanted: SJ4 connector and RV high voltage SJ4 lead (SJ4 system) were implanted in subjects who received a standard of care ICD or CRT-D system for the treatment of heart failure or life-threatening ventricular tachyarrhythmia(s).
Period: Overall Study
Arm/Group | SJ4 System Implanted
Started | 1701 (Total number of subjects consented)
Completed | 866 (Subjects that completed the 60 month follow up visit)
Not Completed | 835
Not completed — Unsuccessful Implant | 4
Not completed — Death | 461
Not completed — Withdrawn - Non-Death | 364
Not completed — Lost to Follow-up | 6

BASELINE CHARACTERISTICS:
Population: Participants had an approved indication, as per ACC/AHA/HRS guidelines, for implantation of an ICD or CRT-D system for treatment of heart failure or life-threatening ventricular tachyarrhythmia(s) and will be implanted with a St. Jude Medical SJ4 system and had given informed consent prior to enrollment.
Arm/Group | SJ4 System Implanted
Number analyzed (Participants) | 1701
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 482
  Male | 1219
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian Or Alaska Native | 1
  Asian | 20
  Black or African American | 235
  Hispanic or Latino | 53
  Iranian | 1
  Middle Eastern | 1
  Native Hawaiian or Pacific Islander | 4
  Other- Non Hispanic | 2
  Persian | 1
  White | 1382
  Hispanic/ Black (Puerto Rican) | 1
Region of Enrollment [Number; unit: participants]
  United States | 1701
New York Heart Association (NYHA) Class [Number; unit: participants] — NHYA classification:Class I-no limitation of physical activity, ordinary physical activity doesn't cause undue breathlessness, fatigue, or palpitations, Class II-slight limitation of physical activity;comfortable at rest; ordinary physical activity results in fatigue, palpitation, dyspnea, Class III-marked limitation of physical activity;comfortable at rest;less than ordinary activity causes fatigue, palpitation, or dyspnea, class IV-Unable to carry on any physical activity without discomfort; symptoms at rest can be present; if any physical activity is undertaken, discomfort is increased.
  participants
    Class 1 | 94
    Class 2 | 541
    Class 3 | 816
    Class 4 | 29
    Not Available | 221
Left Ventricular (LV) Ejection Fraction (%) [Mean (Standard Deviation); unit: Percentage] | 29 (12)
Primary Indication for Device Implant [Number; unit: participants]
  CRT-D Upgrade | 65
  DEFINITE | 5
  Familial Condition | 31
  HF With Wide QRS | 484
  HF Without QRS | 45
  HF Without Sinus Rhythm | 70
  ICD Upgrade | 44
  MADIT II | 228
  PAVE | 14
  Physician Designated | 19
  SCD-HeFT | 409
  Syncope | 39
  VF | 83
  VT | 164
  Not Available | 1

OUTCOME MEASURES:

1. Primary Outcome: Right Ventricle (RV) Bipolar Capture Thresholds
Time Frame: 5 years
Population: Study participants with RV bipolar capture threshold at the 5 year follow up visit.
Measure: Mean (90% Confidence Interval); unit: Volts
Arm/Group | SJ4 System Implanted
Number analyzed (Participants) | 856
Volts | 0.92 [0.89 to 0.95]

2. Primary Outcome: Complication Free Survival Rate Related to the High Voltage RV SJ4 Lead or SJ4 Connector
Time Frame: 5 years
Measure: Number (90% Confidence Interval); unit: percentage of patients
Arm/Group | SJ4 System Implanted
Number analyzed (Participants) | 1701
percentage of patients | 96.4 [95.5 to 97.2]

ADVERSE EVENTS:
Arm/Group | SJ4 System Implanted
Serious Adverse Events (participants affected / at risk) | 0/1701
Other Adverse Events (participants affected / at risk) | 376/1701
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SJ4 System Implanted (N=1701)
RV Lead or DF4 Connector Related Complication (General disorders) | 50 (54) — RV lead or DF4 connector related complications (an adverse event caused by or associated with the study device, system component(s), and or procedure that requires invasive intervention)
System and/or Procedure Related Complication (General disorders) | 44 (64) — Various complications (an adverse event caused by or associated with the study device, system component(s), and or procedure that requires invasive intervention) reported that did not meet the <1% report threshold.
Infection Complication (Infections and infestations) | 36 (37) — Infection complications (an adverse event caused by or associated with the study device, system component(s), and or procedure that requires invasive intervention) reported.
LV Lead Dislodgment or Migration Complication (General disorders) | 21 (24) — LV Lead dislodgement and migration complication (an adverse event caused by or associated with the study device, system component(s), and or procedure that requires invasive intervention).
RA Lead Dislodgement or Migration Complication (General disorders) | 21 (25) — RA lead dislodgement complication (an adverse event caused by or associated with the study device, system component(s), and or procedure that requires invasive intervention).
Lead Dislodgement or Migration <30 days after Implant Complication (Surgical and medical procedures) | 21 (22) — All were resolved with lead repositioning or replacement.
System and/or Procedure Related Observation (General disorders) | 38 (94) — Observations (an adverse event caused by or associated with the study device, system component(s), and or procedure that does not require invasive intervention) that did not meet the <1% reporting threshold.
RV Lead or DF4 Connector Related Observation (General disorders) | 45 (52) — Summary of RV Lead or DF4 Connector Related Observations (an adverse event caused by or associated with the study device, system component(s), and or procedure that does not require invasive intervention).
Elevated LV Pacing Thresholds Observation (General disorders) | 21 (24) — Elevated LV pacing threshold observations ((an adverse event caused by or associated with the study device, system component(s), and or procedure that does not require invasive intervention).
Inappropriate Shock(s) Observation (General disorders) | 33 (36) — Therapy delivered for non-ventricular arrhythmias falling within the VT zones programmed in the device reported observations.
LV Phrenic Nerve/ Diaphragmatic Stimulation Observation (General disorders) | 51 (56) — LV Phrenic nerve/ diaphragmatic stimulation observation(an adverse event caused by or associated with the study device, system component(s), and or procedure that does not require invasive intervention).
RA Oversensing Observation (General disorders) | 40 (47) — RA over sensing observations (an adverse event caused by or associated with the study device, system component(s), and or procedure that does not require invasive intervention).
Bleeding/ Hematoma Observation (Surgical and medical procedures) | 38 (38) — Oozing/bleeding at site of incision following implant/system revision of implanted device system observation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No